CLINICAL TRIAL: NCT05291897
Title: First choIce Antidepressants: General Practitioner's Treatment Approach in the Czech Republic (FIAT)
Brief Title: First choIce Antidepressants: General Practitioner's Treatment Approach in the Czech Republic
Acronym: FIAT
Status: Terminated | Type: Observational
Why Stopped: The number of needed patients wasn't enrolled
Sponsor: Angelini Pharma Česká republika s.r.o. (Industry)
Collaborators: Institut biostatistiky a analýz, s.r.o. (IBA) (Unknown); MINDPAX, s.r.o. (Unknown); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 153(B)LM21212
Record Dates: First submitted 2022-01-12; First posted 2022-03-23 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2022-03

CONDITIONS: Major Depressive Disorder Co-Occurrent With Anxiety; Adult Patients; Newly Diagnosed Depression
Keywords: depression; first choice antidepressant; insomnia; real world data; MDD; MindG bracelets; anxiety; anhedonia; sexual disfunction
MeSH Terms: conditions — Depression; Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Anhedonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
According to the local guidelines (Recommendation for General Practitioners), the first choice Anti-Depressant (AD) in Major Depressive Disorder (MDD) in primary care should be selective serotonin reuptake inhibitors (SSRI), e.g. citalopram, escitalopram, fluoxetine, fluvoxamine, paroxetine, sertraline, in depression with anxiety and insomnia is preferable trazodone and in severer disorders mirtazapine. Despite all these molecules have a very good antidepressant effect, there are differences in side effect scale and tolerability.

The aim of this Study is describing of real treatment practice and MDD management in primary care - aimed to evaluate effectiveness of the treatments in depression and related symptoms: insomnia, anxiety, anhedonia and sexual dysfunction.

The primary objective of the Study is to describe the diagnostic process and treatment patterns in MDD- treatment of choice (pharmacologic with details of first choice antidepressant) in the office of GP's.

The secondary objective is to evaluate efficiency of the treatments in depression and related symptoms: insomnia, anxiety, anhedonia and sexual dysfunction and to monitor the type of side effects and comedication during the 8-weeks treatment.

DETAILED DESCRIPTION:
Research question:

What are the common clinical practices adopted by general practitioner - diagnostic process and treatment of choice (pharmacologic with details of first choice antidepressant) in patients with newly diagnosed depression and how the diagnosis is performed.

Data sources:

Validated questionnaires (PHQ-9, GAD-7, SHAPS), quality of sleep measures with wrist actigraphy monitor. Questions dedicated to sexual dysfunctions. Data about patient's history, diagnosis, treatment and relevant side effects collected directly to the database.

Variables:

Primary Variables Sex and age of the patient. Type of treatment - one of the first line antidepressants available in GP's office (SSRIs, trazodone or mirtazapine) and specifications regarding the treatment approach: initiation dose of treatment, therapeutic dose of treatment, date of the dose increase, total day dose of treatment.

Secondary Variables Insomnia, anxiety and anhedonia will be evaluated by differences of scores of questionnaires (before and after treatment). Sexual dysfunction will be evaluated by differences of answers (before and after treatment).

* Proportional change in total sleep time (TST) before (1 day) /after (8 weeks) the initiation of treatment (TST is defined as the amount of actually sleep time in a sleep episode; this time is equal to the total sleep episode less the awake time).
* Sleep efficiency (time asleep / (total time in bed - time to fall asleep).
* Sleep latency (the duration of time from bedtime, to the onset of sleep).
* Sleep bouts (the number of occurrences of a bout (or multiple bouts), the average length of the bout(s), the total time spent in the bouts, and the total count level of the bouts).
* Sleep fragmentation index (index of restlessness during the sleep period expressed as a percentage).

Monitoring of the type of side effects and comedication during the 8-weeks.

Statistical methods:

Categorical parameters will be described by absolute and relative frequencies. Relative frequencies will be calculated based on the number of patients in relevant subgroup. Continuous parameters will be described by mean and standard deviation (SD) and median with minimum and maximum, together with the total number of non-missing observations.

The differences of the scores of the questionnaires (measured before and after treatment) will be also described by standard characteristics as mean (SD) and median (minimum-maximum). These differences will be tested by paired test (paired t-test or paired Wilcoxon test in dependence on meeting prerequisites). Differences with p-values < 0.05 will be statistically significant (analysis will be performed with level of significance α=0.05).

All statistical tests and confidence intervals will be of exploratory nature.

ELIGIBILITY:
Inclusion Criteria:

* Signing of the Inform Consent Form (Personal Data Protection Consent included)
* Adults male and female newly diagnosed with depression in care of the general practitioner

Exclusion Criteria:

* Patients previously treated with depression or patients treated by a psychiatrist
* Pregnancy and breast-feeding
* Acute myocardial infarction
* Significant risk of suicide
* Concomitant antidepressant medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with newly diagnosed depression included in the Non-Interventional Study (NIS) must be assigned to the therapy before and independently with respect to the decision of being enrolled in the Study.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Description of the type of antidepressant | patient duration: from enrollment to end of treatment for 8 weeks
  The variable type of antidepressant will be observed and evaluated.
Description of the dose of the antidepressant | patient duration: from enrollment to end of treatment for 8 weeks
  The difference between the therapeutic and prescribed dose of antidepressant will be computed as therapeutic dose - prescribed dose.
Description of the increase of dose | patient duration: from enrollment to end of treatment for 8 weeks
  The variable the increase of dose will be computed as changes of dose of comedication drug at the end of follow-up - dose of the drug at the start of follow-up.
Description of the time on an antidepressant without change of dose | patient duration: from enrollment to end of treatment for 8 weeks
  Time on an antidepressant without change of dose will be computed as date of increase of dose - date of enrolment visit.
Description of the maximum daily dose of antidepressant | patient duration: from enrollment to end of treatment for 8 weeks
  The variable maximum total daily dose will be observed and evaluated.

SECONDARY OUTCOMES:
Treatment efficiency - insomnia - change in total sleep time | patient duration: from enrollment to end of treatment for 8 weeks
  Data about insomnia will be collected via a wireless-enabled wrist-worn actigraphy device.
  Variable proportional change in total sleep time is defined as the amount of actual sleep time in a sleep episode; this time is equal to the total sleep episode less the awake time.
Treatment efficiency - insomnia - sleep efficiency | patient duration: from enrollment to end of treatment for 8 weeks
  Data about insomnia will be collected via a wireless-enabled wrist-worn actigraphy device.
  Variable sleep efficiency is defined as time asleep / (total time in bed - time to fall asleep).
Treatment efficiency - insomnia - sleep latency | patient duration: from enrollment to end of treatment for 8 weeks
  Data about insomnia will be collected via a wireless-enabled wrist-worn actigraphy device.
  Variable sleep latency is defined as the duration of time from bedtime, to the onset of sleep.
Treatment efficiency - insomnia - sleep bouts | patient duration: from enrollment to end of treatment for 8 weeks
  Data about insomnia will be collected via a wireless-enabled wrist-worn actigraphy device.
  Variable sleep bouts is defined as the number of occurrences of a bout (or multiple bouts), the average length of the bout(s) will be evaluated and described.
Treatment efficiency - insomnia - sleep bouts | patient duration: from enrollment to end of treatment for 8 weeks
  Data about insomnia will be collected via a wireless-enabled wrist-worn actigraphy device.
  Variable sleep bouts is defined as the number of occurrences of a bout (or multiple bouts), the total time spent in the bouts will be evaluated and described.
Treatment efficiency - insomnia - sleep bouts | patient duration: from enrollment to end of treatment for 8 weeks
  Data about insomnia will be collected via a wireless-enabled wrist-worn actigraphy device.
  Variable sleep bouts is defined as the number of occurrences of a bout (or multiple bouts), the total count level of the bouts will be evaluated and described.
Treatment efficiency - insomnia - sleep fragmentation index | patient duration: from enrollment to end of treatment for 8 weeks
  Data about insomnia will be collected via a wireless-enabled wrist-worn actigraphy device.
  Variable sleep fragmentation index is defined as the index of restlessness during the sleep period expressed as a percentage.
Treatment efficiency - anxiety | patient duration: from enrollment to end of treatment for 8 weeks
  Data about anxiety will be collected via the validated self-administered questionnaire - Generalized Anxiety Disorder Questionnaire (GAD-7). Differences in the score of the questionnaire (measured before and after treatment) will be computed as the score of the questionnaire after treatment - the score of the questionnaire before treatment.
  Scale values:
  GAD-7 - total scores ranged from 0 to 21. A higher total GAD-7 score indicated higher levels of the present state of anxiety.
Treatment efficiency - anhedonia | patient duration: from enrollment to end of treatment for 8 weeks
  Data about anhedonia will be collected via the validated self-administered questionnaire - Snaith-Hamilton Pleasure Scale (SHAPS). Differences in the score of the questionnaires (measured before and after treatment) will be computed as the score of the questionnaire after treatment - the score of the questionnaire before treatment.
  Scale values:
  SHAPS - total scores ranged from 0 to 14. A higher total SHAPS score indicated higher levels of the present state of anhedonia.
Treatment efficiency - level of depression | patient duration: from enrollment to end of treatment for 8 weeks
  Data will be collected via the validated self-administered questionnaire-Patient Health Questionnaire-9 (PHQ-9) - Patient Health Questionnaire. Differences in the score of the questionnaire (measured before and after treatment) will be computed as the score of the questionnaire after treatment - the score of the questionnaire before treatment.
  Scale values:
  PHQ-9 - total scores ranged from 0 to 27. A higher total PHQ-9 score indicated higher levels of the present state of depression.
Treatment efficiency - sexual dysfunction | patient duration: from enrollment to end of treatment for 8 weeks
  Sexual dysfunction data will be collected via dedicated questions. Answers to questions about sexual dysfunction at the start and end of treatment will be compared and evaluated.
Treatment efficiency - adverse events | patient duration: from enrollment to end of treatment for 8 weeks
  Monitoring of the type of side effects during the 8-weeks. The summary of Adverse events (AE) / Severe Adverse Events (SAE) will present the number and percentage of patients who had at least one AE. The data on AEs/SAEs will be listed.
Monitoring of the type of comedication during the 8-weeks | patient duration: from enrollment to end of treatment for 8 weeks
  Monitoring of the comedication during the 8-weeks. Changes in comedications between the initial and terminal visits will be evaluated and described.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Španiel, MD, PhD, Principal Investigator — National Institute of Mental Health (NIMH)
Locations (6):
- Czechia (6):
  - MUDr. František Rolinek, s.r.o., Brno
  - Artemisia všeobecné lékařství, s.r.o., Brno
  - MEDIGATE Care s.r.o., Hradec Králové
  - AAAmbulance, s.r.o., Litoměřice
  - Poliklinika Prosek, Prague
  - PragMed, s.r.o., Prague